CLINICAL TRIAL: NCT05277961
Title: Quantification of DNA Repair Products in the Urine After Ultraviolet Radiation of the Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Sygehus Lillebaelt (Other)
Responsible Party: Principal Investigator, Catharina Margrethe Lerche, Associate Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-20076172
Record Dates: First submitted 2022-02-17; First posted 2022-03-14 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Ultraviolet Rays; Injury; DNA Adduct Formation; DNA Damage, Radiation Induced; DNA Damage
Keywords: DNA repair; DNA damage; Thymine dimer; Ultraviolet radiation; Urine; HPLC-MS
MeSH Terms: conditions — Wounds and Injuries | interventions — Ultraviolet Rays

STUDY DESIGN:
Intervention Model Description: Two groups of healthy volunteers are UV radiated with two different dosage regimen.
  DNA repair excreted in the urine are quantified by LC-MS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UVR Dose 1x3SED (Experimental): UVR Dose 1x3 standard erytheme dose (SED)
  Interventions: Radiation: Ultraviolet radiation
- UVR dose 3x1SED (Experimental): UVR dose 3x1 standard erythema dose (SED)
  Interventions: Radiation: Ultraviolet radiation

INTERVENTIONS:
Radiation: Ultraviolet radiation — UV6 tubes

SUMMARY:
Purpose of the experiment The investigators know that DNA damage is formed in the skin by sun exposure of the thymine-dimer type. Many of these injuries are repaired and excreted through the urine.

The purpose of the study is to quantify DNA damage in the urine after ultraviolet (UV) irradiation of the skin in healthy subjects. The investigators would like to investigate which day after two different irradiation regimens the highest secretion of thymine dimers occurs. If the investigators establish such a test system, it will be possible to test potential photoprotective substances or potential photocarcinogenic substances.

Method of the experiment, design, and examination procedures The subjects (n = 16-20) are recruited by a post on Bispebjerg's hospital website. Based on this, subjects are divided into 2 groups of 8-10 people. Group 1 is irradiated 3 times with 1 standard erythema dose (SED). 1 SED corresponds to approx. 10 minutes sun around 13 pm on a good Danish summer day. Group 2 is irradiated once with 3 SED, which corresponds to approx. 30 minutes around 13 pm on a good Danish summer day. The irradiation is carried out on day 1 for group 2 and days 1, 2 and 3 for group 1.

Subjects are irradiated in a full-body UV cabin (Waldmann, Willing-Schwenningen, Germany) with 26 F85 / 100W UV6 tubes (290-350 nm, broad-spectrum). 13 seconds of illumination, equivalent to 1 SED. The subjects are standing in the cabin and have a screen on so that their eyes and face are not exposed to radiation. When irradiated, the subjects must only wear underwear, which for men are underpants/boxer shorts, while for women it is bras and panties. The experiment is performed between October and March, to avoid that the subjects do not simultaneously receive UV radiation from the sun and thus form DNA damage.

Subjects must collect morning urine in dispensed containers and must store it in their own freezer until the final visit. Morning urine (2x 50 mL) is collected before irradiation, called day 1, and even until day 8 after the last exposure, ie. day 10 for group 1 and day 8 for group 2. Before the first exposure, pigment and redness are measured on the subjects. Pigment and redness measurements are performed on the back, chest, and shoulder.

DETAILED DESCRIPTION:
Project title:

Determination of DNA repair products in urine after UV irradiation of the skin

1. Purpose

   Problem definition

   DNA damage is formed in the skin by sun exposure. The most common DNA damage is called thymine dimers. Many of these injuries are repaired by "Nucleotide excision repair" (NER) and excreted through the urine. The importance of this repair mechanism is seen in patients with defects in their NER, who have a very high risk of developing skin cancer. The investigators want to be able to quantify the amount of thymine dimers in the urine after ultraviolet (UV) irradiation of the skin. With the establishment of such a test system, it will eventually be possible to test potential photoprotective substances or potential photocarcinogenic substances based on damage measured in the urine after a known UV dose. The investigators would like to investigate when the highest secretion of this type of DNA damage occurs using two different irradiation regimens. It has previously been possible to quantify thymine dimers in the urine using an isotope method, but that method is no longer available and it is desirable to avoid isotopes. The investigators have developed a new method based on Ultra High-pressure Liquid Chromatography-Mass Spectrometry (UHPLC-MS).

   Hypothesis

   The investigators have the hypothesis that maximum excretion of thymine dimers in the urine occurs 1-4 days after UV irradiation of the skin.

   Background

   Ultraviolet (UV) radiation causes DNA damage in the skin that can eventually lead to skin cancer. Thymine dimer is a DNA damage that is only formed when UV rays hit DNA in the skin cells. Nucleotide excision repair (NER) repairs and removes thymine dimers in the individual cell, which are then excreted in the urine. Thymine dimers in the urine are a biomarker for total DNA repair. In the past, a method for quantifying thymine dimers in urine using isotope labeling has existed. The method was very sensitive but had a long analysis time and in addition, it is an advantage from a work environment to avoid working with radioactive isotopes.

   The investigators have succeeded in developing a new method of analysis using UHPLC-MS. This method has high sensitivity and high selectivity while having a fast analysis time. In addition, this equipment is capable of analyzing multiple DNA modifications. Furthermore, there is high sensitivity and high selectivity. This study is a proof-of-concept study in which the investigators would like to investigate when the most optimal time for urine collection is after two different irradiation regimens. The perspective is to be able to use the method to find new potential photo-protective as well as photocarcinogenic substances.
2. Method

   Study design for healthy subjects

   The subjects (n = 16-20) are recruited by a notice on Bispebjerg's hospital website. Subjects will be invited to an initial screening visit where participants will receive oral information about the study by trial supervisor Catharina Lerche. The meeting takes place in a separate room to ensure a safe and quiet environment. Subjects will be informed that participants can bring an assistant if wished. Written informed consent will be ensured, and takes place at least 24 hours after the screening visit.

   Based on this, subjects are divided into 2 groups of 8-10 people. Group 1 is irradiated 3 times with 1 standard erythema dose (SED). 1 SED corresponds to approx. 10 min sun around kl. 13 on a good Danish summer day. Group 2 is irradiated once with 3 SED, which corresponds to approx. 30 min around kl. 13 on a good Danish summer day. The irradiation is carried out on day 1 for group 2 and days 1, 2, and 3 for group 1.

   Subjects are irradiated in a full-body UV cabin (Waldmann, Willing-Schwenningen, Germany) with 26 F85 / 100W UV6 tubes (290-350 nm, broad-spectrum). The irradiation time is set on a timer clock so that the UV cabin switches off after the desired irradiation time. The irradiation time is 16 seconds for a 1 SED and 43 seconds for a 3 SED. The UV cabin is measured using calibrated equipment, which is also used to measure UV cabins in the clinic, which are used for patients. The subjects stand up in the cabin and have a screen on so that their eyes and face are not exposed to radiation. When lighting, subjects should only wear underwear, which for men are underpants/boxer shorts, while for women it is bras and panties. The experiment is performed between October and March, to avoid that the subjects do not simultaneously receive UV radiation from the sun and thus can form DNA damage. Subjects must collect morning urine in dispensed containers and must store it in their own freezer until the final visit.

   Morning urine (2x 50 ml) is collected before irradiation, called day 1 and even until day 8 after the last irradiation, ie. day 10 for group 1 and day 8 for group 2. 2 x 50 ml x 10 in total 1000 ml of urine are collected for group 1 and 2 x 50 ml x 8 a total of 800 ml of urine for group 2. Before and after each illumination are measured pigment and redness on the subjects as well as on final visits. Pigment and redness measurements are performed on the back, chest, and buttocks.
3. Statistical considerations

   Previous studies have observed an increase of 1.7 nmol with a scattering (SD) of 1.3 nmol 4, power of 0.80, as well as significance level of 0.05 in a paired test, then 7 people must complete the study when the investigators set the power to 0.80 and have a significance level of 0.05 and use the paired test (Power and Sample Size Calculation, PS, Vanderbilt University; version 3.1.2). As the study lasts up to 10 days, dropouts can be expected, and therefore 8-10 are included in each of the two groups, ie. a total of 16-20 healthy subjects.
4. Risks, side effects, and disadvantages in the short and long term

   There is a slight risk of short-term redness after lighting, as well as after staying in the sun. The UV doses (3 SED) have been chosen so that almost all Danes will avoid redness. The total UV dose corresponds to a ½ hour stay in the sun in the middle of the day during the summer in Denmark. All subjects will be informed both orally and in writing about the risks and possible side effects.

   No biobank will be created. The urine samples are analyzed immediately after collection. Excess biological material is destroyed immediately after analysis.
5. Quality control

   The Helsinki II Declaration will be respected as well as the standards of good clinical research. Respect for privacy as well as for physical and mental integrity in patients is maintained. The study will be registered at the Knowledge Center for Data Reporting, the Capital Region, in the electronic system Pactius.
6. Data protection and storage The general data protection regulation will be respected. Research using data from the capital region is considered public research. The use and distribution of data collected in this study will be discussed with patients during the consent process. The project is reported to the Knowledge Center for Data Reporting, the Capital Region of Denmark in the electronic system Pactius. A list of the subjects' names, study ID, and date of birth is prepared. All collected data will be anonymised and protected by Danish legislation regarding the handling of personal data and the Health Act. Data are registered and stored for 5 years after completion of the study at the Department of Dermatology, Bispebjerg Hospital.
7. Economy It is Pharmacist Catharina Lerche, Professor Hans Christian Wulf, and Engineer Peter Philipsen who have taken the initiative for the experiment, and the investigators are all paid by the skin department, Bispebjerg hospital. There are no contributions from companies or external funds to this experiment.
8. Information for subjects The principal investigator, Catharina M. Lerche, is responsible for providing clear oral and written information about the goals, designs, and risks of the study, as stated in "Information and consent to participate in health science research projects" by the Ministry of Health and the Elderly. In undisturbed surroundings, the participant will be made aware of their right to have one / or more attendants present, that participation is voluntary and that withdrawal is possible at any time during the study. Subjects are given sufficient reflection time (at least 24 hours). Subjects will be asked to sign a consent form.
9. Publication of results Positive, negative, and conclusive results will be published. The aim is to publish and present the results in a peer-reviewed international dermatology journal and/or at dermatological conferences. The intellectual property rights to the results belong to Bispebjerg Hospital. Publications will comply with the Vancouver Guidelines.
10. Ethics Personal information and urine samples are processed in accordance with the Personal Data Act and the Health Act. The project is also implemented with minimal health and safety risks for the participants. It is expected that the potential risks of adverse effects in this study are very small. The potential for evidence-based future gains and the future perspectives that this study may provide should be weighed against trial participation. Danish laws on patients' rights and compensation are followed.

ELIGIBILITY:
Inclusion criteria:

* Over the age of 18
* Written informed consent from the subject

Exclusion criteria:

* Immunosuppressed individuals
* Sun holiday/ski holiday/solarium 4 weeks before the trial starts
* Skin disease
* Medicines that cause photosensitivity or affect DNA repair
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Determination of days where the concentration of excreted thymine dimers (a marker of DNA damage) is the highest in the urine after UVR exposure of the skin. | 10 days
  Each participant of group 1 will provide a total of 1000 ml (2 x50 ml x10 days) of urine and participants of group 2 will provide a total of 800 ml (2 x 50 ml x 8 days) of urine at the end of the experiment. UVR induced thymine dimers repaired and excreted in the urine will be quantified (by Ultra High-pressure Liquid Chromatography-Mass Spectrometry (UHPLC-MS) from urine collected before and after irradiation regimes. The highest concentration of thymine dimers in urine will indicate the most optimal time for urine collection after irradiation.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Christian Wulf, PhD, Study Chair — RegionH
Locations (1):
- Bispebjerg Hospital, Department of Dermatology, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brash DE, Rudolph JA, Simon JA, Lin A, McKenna GJ, Baden HP, Halperin AJ, Ponten J. A role for sunlight in skin cancer: UV-induced p53 mutations in squamous cell carcinoma. Proc Natl Acad Sci U S A. 1991 Nov 15;88(22):10124-8. doi: 10.1073/pnas.88.22.10124. PMID 1946433
- [Background] Martens MC, Emmert S, Boeckmann L. Sunlight, Vitamin D, and Xeroderma Pigmentosum. Adv Exp Med Biol. 2020;1268:319-331. doi: 10.1007/978-3-030-46227-7_16. PMID 32918226
- [Background] Le Curieux F, Hemminki K. Cyclobutane thymidine dimers are present in human urine following sun exposure: quantitation using 32P-postlabeling and high-performance liquid chromatography. J Invest Dermatol. 2001 Aug;117(2):263-8. doi: 10.1046/j.1523-1747.2001.01416.x. PMID 11511303
- [Background] Petersen B, Wulf HC, Triguero-Mas M, Philipsen PA, Thieden E, Olsen P, Heydenreich J, Dadvand P, Basagana X, Liljendahl TS, Harrison GI, Segerback D, Schmalwieser AW, Young AR, Nieuwenhuijsen MJ. Sun and ski holidays improve vitamin D status, but are associated with high levels of DNA damage. J Invest Dermatol. 2014 Nov;134(11):2806-2813. doi: 10.1038/jid.2014.223. Epub 2014 May 20. PMID 24844860

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT05277961/Prot_SAP_002.pdf
  • Informed Consent Form (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT05277961/ICF_001.pdf